CLINICAL TRIAL: NCT06766929
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VSA012 After Single Ascending Doses in Healthy Volunteers
Brief Title: A Phase I Clinical Study of VSA012 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Visirna Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSA012-1001
Record Dates: First submitted 2024-12-29; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VSA012 (Experimental): Single ascending doses of VSA012
  Interventions: Drug: VSA012
- Placebo (Placebo Comparator): Single ascending doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSA012 — subcutaneous injection
  Arms: VSA012
Drug: Placebo — subcutaneous injection
  Arms: Placebo

SUMMARY:
The complement system is an important component of the innate immune system. Abnormal activation, inadequate regulation and control of the complement system, as well as impaired and dysfunctional effector functions, underlie complement mediated diseases. VSA012 targeting complement system has the potential to treat a variety of diseases associated with abnormal activation of the complement system (e.g. PNH) .The purpose of VSA012-1001 is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of VSA012 Injection in adult healthy volunteers (HVs). HVs will receive a single dose of VSA012 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent and to comply with study requirements
* Participants must be non-pregnant/non-lactating
* Healthy volunteers must be willing to be vaccinated with a meningococcal and pneumococcal vaccine.
* Body Mass Index (BMI) between 18.0 and 30.0 kg/m2
* No abnormal finding of clinical relevance at the Screening evaluation that, in the opinion of the Investigator, could adversely impact participant safety or adversely impact study results.

Exclusion Criteria:

* History of recurrent or chronic infections including infections caused by encapsulated bacterial organisms or viruses
* History of active bacterial, viral, or fungal infection within 14 days prior to treatment administrations
* Seropositive for Human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* History of meningococcal infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (AEs) and/or Serious Adverse Events (SAEs) | up to Day 180

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of VSA012: Maximum Observed Plasma Concentration (Cmax) | Up to 48 hours post-dose
PK of VSA012: Time to Maximum Observed Plasma Concentration (Tmax) | Up to 48 hours post-dose
PK of VSA012: Area Under the Plasma Concentration Versus Time Curve | Up to 48 hours post-dose
Change from Baseline in Serum Complement Factor B (CFB) | Up to Day 180
Change from Baseline in Serum Complement Alternative Pathway (CAP) | up to Day 180
The incidence of ADA | up to Day 180

IPD SHARING:
Plan to Share IPD: No